CLINICAL TRIAL: NCT02692027
Title: Same Day Community-based ART Initiation Versus Clinic-based Pre-ART Assessment and Counselling for Individuals Newly Tested HIV-positive During Community-based HIV Testing in Rural Lesotho - a Randomized Controlled Trial
Brief Title: Same-day ART Initiation Versus Standard of Care After Positive HIV-test Result in Rural Lesotho
Acronym: CASCADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: SolidarMed - Swiss Organization for Health in Africa (Unknown); Ministry of Health, Lesotho (Other Government); District Health Management Team of Butha-Buthe, Lesotho (Other); University of Basel (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Niklaus Labhardt, MD, MIH, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CASCADE
Record Dates: First submitted 2016-02-21; First posted 2016-02-25 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: HIV Infection
Keywords: Community-based initiation of antiretroviral therapy; Home-based HIV testing and counseling; Lesotho; Sub-sahara Africa; antiretroviral therapy; AIDS; Test and treat
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): Standard of care in Lesotho. ART-initiation after at least two clinic visits for pre-ART counseling and monthly follow-up visits at the clinic thereafter.
  Interventions: Other: Standard of care
- Same-day ART initiation with less frequent follow-up visits (Experimental): Proposition of same-day ART initiation with less frequent follow-up visits thereafter.
  Interventions: Other: Same-day ART initiation

INTERVENTIONS:
Other: Same-day ART initiation — Participants tested HIV-positive during community-based HIV testing and randomized to the intervention group receive post-test counseling and on-the-spot clinical and laboratory assessment. Directly after the positive HIV-test result the study nurse assesses the participant clinically and performs point-of-care laboratory baseline testing. Thereafter, the participant receives a standardized short adherence counselling. After adherence counseling the participant is offered to start ART immediately. Those who decide to start ART during the visit or intend to start within seven days will receive a 30 day ART-supply and an follow-up appointment at the clinic within 12 to 16 days.
  In order to reduce travel time and transport cost, participants who are clinically stable, will have their follow-up visits and ART refills more widely spaced with appointments at 6 weeks, 3, 6, (9) and 12 months after ART initiation.
  Arms: Same-day ART initiation with less frequent follow-up visits
Other: Standard of care — Individuals found HIV-positive during the community-based HIV testing campaigns and randomized to the control arm receive post-test counselling and a referral letter with an appointment at their chosen health facility. On the first visit to the clinic, the participant receives laboratory assessment and a first adherence counselling session. The participant must then return to the clinic to receive his/her laboratory results and to undergo a second adherence counselling session.
  Once the participant has started ART, the first and second follow-up visits are scheduled for 14 and 28 days after ART initiation, respectively. Thereafter, follow-up visits are scheduled monthly until 6 months after ART initiation. If the participant is clinically stable, clinical follow-up visits may then be spaced to 3-monthly intervals, but refills of ART must still be collected on a monthly basis.
  Arms: Standard of care

SUMMARY:
The CASCADE-trial is a two-armed open-label randomized controlled trial conducted in rural Lesotho. Participants who were tested HIV-positive during community-based HIV testing and counseling campaigns are randomized to the intervention or control arm. Allocation is 1:1 with parallel assignment.

Participants in the control arm follow the standard of care after a community-based HIV test result: They are referred to the nearest clinic where they will receive baseline laboratory testing and adherence counseling. After at least 2 clinic visits for adherence counseling they can start anti-retroviral therapy (ART). After ART-initiation they have to attend monthly follow-up at the clinic for drug refill. Individuals randomized to the intervention arm are proposed same day community-based ART initiation combined with less frequent follow-up visits. The primary outcomes are linkage to care at 3 months and viral suppression at 12 months after having tested HIV-positive during the community-based HIV testing and counseling campaigns.

DETAILED DESCRIPTION:
A published version of the trial protocol can be downloaded at:

http://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-016-2972-6

Background

In November 2014 the Joint United Nations Programme on HIV/AIDS (UNAIDS) published the 90-90-90 targets for 2020 (UNAIDS 2014). The strategy aims at a massive scale-up in coverage of antiretroviral therapy (ART) among individuals infected with HIV. Based on accumulated evidence that viral suppression through successful ART reduces the risk of transmission(Cohen 2011), it is expected that - if achieved - the 90-90-90 targets would lead to a reduction of the yearly global HIV-incidence from 2 million currently to 500'000 by 2020 (Jones 2014). In 2015 two randomized controlled trials showed the benefit of starting ART as early as possible for infected individuals - even if CD4-cell counts were above the threshold of 500 cells/mL (TEMPRANO 2015; INSIGHT START 2015), leading the World Health Organization (WHO) to recommend that anyone infected with HIV should start ART as soon as possible after diagnosis (WHO 2015). A "seek-test-treat" strategy bears, however, unprecedented challenges in settings where HIV is hyperendemic and resources may be limited (Hull 2014; Delva 2015).

The Continuum of Care Cascade ("the cascade") involves the steps HIV-infected individuals have to take in order to achieve viral suppression. It starts with knowing one's HIV status, continues with linkage to care after a positive HIV test, initiation of ART, uninterrupted continuation of ART (retention in care and adherence to medication), and ends with viral suppression (MacCarthy 2015). Already prior to announcement of the "seek-test-and-treat" approach, weaknesses in the cascade often hampered the effectiveness of HIV programs in resource-rich as well as resource-poor settings (Yehia 2015; Kratzer 2012). In Sub-Saharan Africa the care cascade is still far from the 90-90-90 targets with only 29% of infected individuals estimated to be on ART and virally suppressed in 2013. In order to achieve the UNAIDS targets innovative, effective, and practical approaches for improving the care cascade are thus urgently needed (Mills 2013; Piot 2015).

Linkage to care after an initial positive HIV test has been described as the "Achilles' heel" of the care cascade (Nachega 2014). Most studies from Sub-Saharan Africa report linkage rates lower than 50% (Naik 2015; Parker 2015; Clouse 2013; Gerdts 2014). In a cluster-randomized trial comparing home-based with mobile-clinic HIV testing and counselling (HTC) in Lesotho, only 25% of newly tested HIV-positive individuals accessed care within one month after the test (Labhardt 2014).

Several interventions have been shown to improve linkage to care, such as point-of-care CD4 count directly after a positive HIV test, immediate start of cotrimoxazole prophylaxis, incentives such as food-assistance, extended post-test counselling during home-visits, or community-workers accompaniment. However, controlled studies testing programmatic intervention packages for improving linkage to care are still largely lacking (Okeke 2014; Govindasamy 2014). Furthermore, it must be noted that interventions, such as patient-accompaniment or food support are resource intensive and may work in small NGO-driven projects, but are not sustainable on a larger scale (Posse 2013). In a systematic review addressing barriers for linkage to care, transport cost and distance were the most frequently cited factors for patients not enrolling in care after a positive HIV test (Govindasamy 2012).

Objective of the trial

This CASCADE trial tests the effectiveness of same day home-based ART initiation after a positive HIV test in combination with a reduction of the frequency of follow-up visits to the clinic as a pragmatic and programmatically feasible approach to improve linkage to care, retention in care, and viral suppression.

It is a two-armed open-label randomized controlled trial. Allocation is 1:1 with parallel assignment. The intervention is targeted to individuals who tested HIV-positive during community-based HTC.

Recruitment and participants

Participants will be recruited during community-based HTC campaigns in the district of Butha-Buthe, in northern Lesotho. Home-based HTC campaigns will be conducted for an anticipated period of 3 months beginning at the end of February in the catchment areas of six health care facilities - four nurse-led health centers, one missionary and one public hospital.

Three teams consisting of 4 lay counsellors, each supervised by one professional counsellor and a nurse visit all households in randomly pre-selected areas proposing HTC to all household members. If a household member tests HIV positive during the HTC campaign and eligible for the CASCADE trial, he/she will be randomized to one of the two arms.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection newly diagnosed during community-based HTC-campaigns
* Never been on triple-ART
* Lives and/or works in the district of Butha-Buthe and declares to seek follow-up at one of the 6 health facilities involved in the study
* Signed written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding
* Already enrolled in chronic care for another disease, such as tuberculosis or diabetes
* Clinical WHO-stage 4 or active tuberculosis
* Positive cryptococcal antigen test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Linkage to care | 90 days
  Linkage to care within 3 months after having been tested HIV positive during the HTC-campaign. A patient is considered to have linked to care if he/she attends the clinic at least once within 90 days after HIV diagnosis.
Viral suppression | 12 months
  Viral suppression 12 months after positive HIV test result. Viral suppression is defined as a viral load <100 copies/mL between 11 and 14 months after diagnosis of HIV-infection.

SECONDARY OUTCOMES:
1-year retention in care | 12 months
  Proportion confirmed dead (death record at clinic or confirmed by a first-grade relative), lost to follow-up (not attending the clinic 11-14 months after HIV-test and not confirmed dead), and retained in care (on ART, attends the clinic)
Viral suppression under ART | 6 months after ART initiation
  Viral load <100 copies/mL among those who started ART 5-7 months after ART-initiation.
Change in body weight | 12 months
Change in CD4 cell count | 12 months
Change in haemoglobin | 12 months
New clinical WHO stage 3 or 4 events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus D Labhardt, MD, MIH, Principal Investigator — Swiss Tropical & Public Health Institute; Tracy R Glass, PhD, Study Chair — Swiss Tropical & Public Health Institute
Locations (1):
- Butha-Buthe District Hospital, Butha-Buthe, Lesotho

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 90-90-90 An ambitious treatment target to help end the AIDS epidemic. UNAIDS / JC2684 (accessed October 30th 2014 at www.unaids.org) 2014.
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] INSIGHT START Study Group; Lundgren JD, Babiker AG, Gordin F, Emery S, Grund B, Sharma S, Avihingsanon A, Cooper DA, Fatkenheuer G, Llibre JM, Molina JM, Munderi P, Schechter M, Wood R, Klingman KL, Collins S, Lane HC, Phillips AN, Neaton JD. Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection. N Engl J Med. 2015 Aug 27;373(9):795-807. doi: 10.1056/NEJMoa1506816. Epub 2015 Jul 20. PMID 26192873
- [Background] Jones A, Cremin I, Abdullah F, Idoko J, Cherutich P, Kilonzo N, Rees H, Hallett T, O'Reilly K, Koechlin F, Schwartlander B, de Zalduondo B, Kim S, Jay J, Huh J, Piot P, Dybul M. Transformation of HIV from pandemic to low-endemic levels: a public health approach to combination prevention. Lancet. 2014 Jul 19;384(9939):272-9. doi: 10.1016/S0140-6736(13)62230-8. Epub 2014 Apr 14. PMID 24740087
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] Hull M, Lange J, Montaner JS. Treatment as prevention--where next? Curr HIV/AIDS Rep. 2014 Dec;11(4):496-504. doi: 10.1007/s11904-014-0237-5. PMID 25384357
- [Background] Delva W, Abdool Karim Q. The HIV epidemic in Southern Africa - Is an AIDS-free generation possible? Curr HIV/AIDS Rep. 2014 Jun;11(2):99-108. doi: 10.1007/s11904-014-0205-0. PMID 24676559
- [Background] MacCarthy S, Hoffmann M, Ferguson L, Nunn A, Irvin R, Bangsberg D, Gruskin S, Dourado I. The HIV care cascade: models, measures and moving forward. J Int AIDS Soc. 2015 Mar 2;18(1):19395. doi: 10.7448/IAS.18.1.19395. eCollection 2015. PMID 25735869
- [Background] Yehia BR, Stephens-Shields AJ, Fleishman JA, Berry SA, Agwu AL, Metlay JP, Moore RD, Christopher Mathews W, Nijhawan A, Rutstein R, Gaur AH, Gebo KA; HIV Research Network. The HIV Care Continuum: Changes over Time in Retention in Care and Viral Suppression. PLoS One. 2015 Jun 18;10(6):e0129376. doi: 10.1371/journal.pone.0129376. eCollection 2015. PMID 26086089
- [Background] Kranzer K, Govindasamy D, Ford N, Johnston V, Lawn SD. Quantifying and addressing losses along the continuum of care for people living with HIV infection in sub-Saharan Africa: a systematic review. J Int AIDS Soc. 2012 Nov 19;15(2):17383. doi: 10.7448/IAS.15.2.17383. PMID 23199799
- [Background] Mills EJ, Nachega JB, Ford N. Can we stop AIDS with antiretroviral-based treatment as prevention? Glob Health Sci Pract. 2013 Mar 21;1(1):29-34. doi: 10.9745/GHSP-D-12-00053. eCollection 2013 Mar. PMID 25276515
- [Background] Piot P, Abdool Karim SS, Hecht R, Legido-Quigley H, Buse K, Stover J, Resch S, Ryckman T, Mogedal S, Dybul M, Goosby E, Watts C, Kilonzo N, McManus J, Sidibe M; UNAIDS-Lancet Commission. Defeating AIDS--advancing global health. Lancet. 2015 Jul 11;386(9989):171-218. doi: 10.1016/S0140-6736(15)60658-4. Epub 2015 Jun 24. No abstract available. PMID 26117719
- [Background] Nachega JB, Uthman OA, del Rio C, Mugavero MJ, Rees H, Mills EJ. Addressing the Achilles' heel in the HIV care continuum for the success of a test-and-treat strategy to achieve an AIDS-free generation. Clin Infect Dis. 2014 Jul;59 Suppl 1(Suppl 1):S21-7. doi: 10.1093/cid/ciu299. PMID 24926028
- [Background] Naik R, Doherty T, Jackson D, Tabana H, Swanevelder S, Thea DM, Feeley FG, Fox MP. Linkage to care following a home-based HIV counselling and testing intervention in rural South Africa. J Int AIDS Soc. 2015 Jun 8;18(1):19843. doi: 10.7448/IAS.18.1.19843. eCollection 2015. PMID 26058983
- [Background] Parker LA, Jobanputra K, Rusike L, Mazibuko S, Okello V, Kerschberger B, Jouquet G, Cyr J, Teck R. Feasibility and effectiveness of two community-based HIV testing models in rural Swaziland. Trop Med Int Health. 2015 Jul;20(7):893-902. doi: 10.1111/tmi.12501. Epub 2015 Apr 2. PMID 25753897
- [Background] Clouse K, Pettifor AE, Maskew M, Bassett J, Van Rie A, Behets F, Gay C, Sanne I, Fox MP. Patient retention from HIV diagnosis through one year on antiretroviral therapy at a primary health care clinic in Johannesburg, South Africa. J Acquir Immune Defic Syndr. 2013 Feb 1;62(2):e39-46. doi: 10.1097/QAI.0b013e318273ac48. PMID 23011400
- [Background] Gerdts SE, Wagenaar BH, Micek MA, Farquhar C, Kariaganis M, Amos J, Gimbel S, Pfeiffer J, Gloyd S, Sherr K. Linkage to HIV care and antiretroviral therapy by HIV testing service type in Central Mozambique: a retrospective cohort study. J Acquir Immune Defic Syndr. 2014 Jun 1;66(2):e37-44. doi: 10.1097/QAI.0000000000000081. PMID 24326605
- [Background] Labhardt ND, Motlomelo M, Cerutti B, Pfeiffer K, Kamele M, Hobbins MA, Ehmer J. Home-based versus mobile clinic HIV testing and counseling in rural Lesotho: a cluster-randomized trial. PLoS Med. 2014 Dec 16;11(12):e1001768. doi: 10.1371/journal.pmed.1001768. eCollection 2014 Dec. PMID 25513807
- [Background] Okeke NL, Ostermann J, Thielman NM. Enhancing linkage and retention in HIV care: a review of interventions for highly resourced and resource-poor settings. Curr HIV/AIDS Rep. 2014 Dec;11(4):376-92. doi: 10.1007/s11904-014-0233-9. PMID 25323298
- [Background] Govindasamy D, Meghij J, Kebede Negussi E, Clare Baggaley R, Ford N, Kranzer K. Interventions to improve or facilitate linkage to or retention in pre-ART (HIV) care and initiation of ART in low- and middle-income settings--a systematic review. J Int AIDS Soc. 2014 Aug 1;17(1):19032. doi: 10.7448/IAS.17.1.19032. eCollection 2014. PMID 25095831
- [Background] Posse M, Baltussen R. Costs of providing food assistance to HIV/AIDS patients in Sofala province, Mozambique: a retrospective analysis. Cost Eff Resour Alloc. 2013 Aug 28;11(1):20. doi: 10.1186/1478-7547-11-20. PMID 24103560
- [Background] Govindasamy D, Ford N, Kranzer K. Risk factors, barriers and facilitators for linkage to antiretroviral therapy care: a systematic review. AIDS. 2012 Oct 23;26(16):2059-67. doi: 10.1097/QAD.0b013e3283578b9b. PMID 22781227
- [Derived] Amstutz A, Brown JA, Ringera I, Muhairwe J, Lejone TI, Klimkait T, Glass TR, Labhardt ND. Engagement in Care, Viral Suppression, Drug Resistance, and Reasons for Nonengagement After Home-Based Same-Day Antiretroviral Therapy Initiation in Lesotho: A Two-Year Follow-up of the CASCADE Trial. Clin Infect Dis. 2020 Dec 17;71(10):2608-2614. doi: 10.1093/cid/ciz1126. PMID 31781759
- [Derived] Labhardt ND, Ringera I, Lejone TI, Amstutz A, Klimkait T, Muhairwe J, Glass TR. Effect and cost of two successive home visits to increase HIV testing coverage: a prospective study in Lesotho, Southern Africa. BMC Public Health. 2019 Nov 1;19(1):1441. doi: 10.1186/s12889-019-7784-z. PMID 31676001
- [Derived] Labhardt ND, Ringera I, Lejone TI, Klimkait T, Muhairwe J, Amstutz A, Glass TR. Effect of Offering Same-Day ART vs Usual Health Facility Referral During Home-Based HIV Testing on Linkage to Care and Viral Suppression Among Adults With HIV in Lesotho: The CASCADE Randomized Clinical Trial. JAMA. 2018 Mar 20;319(11):1103-1112. doi: 10.1001/jama.2018.1818. PMID 29509839
- [Derived] Labhardt ND, Ringera I, Lejone TI, Masethothi P, Thaanyane T, Kamele M, Gupta RS, Thin K, Cerutti B, Klimkait T, Fritz C, Glass TR. Same day ART initiation versus clinic-based pre-ART assessment and counselling for individuals newly tested HIV-positive during community-based HIV testing in rural Lesotho - a randomized controlled trial (CASCADE trial). BMC Public Health. 2016 Apr 14;16:329. doi: 10.1186/s12889-016-2972-6. PMID 27080120